CLINICAL TRIAL: NCT07216755
Title: Impact of Respiratory Muscle Training and Nitrate Therapy on Exercise Tolerance in Simulated Altitude
Brief Title: Effects of Breathing Training and Nitrate on Exercise at Simulated Altitude
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Embry-Riddle Aeronautical University (Other)
Responsible Party: Principal Investigator, Scott Kohman Ferguson, Assistant Professor, Embry-Riddle Aeronautical University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 25-077; 1R15HL173855-01A1 (NIH)
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adults; Mechanical Ventilation Dependence; Hypoxia; Exercise Training; Exercise Intolerance; Dietary Supplement; Nitrate Supplementation; Inspiratory Muscle Training
MeSH Terms: conditions — Hypoxia | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RMT + Nitrate Supplementation (Experimental): Participants complete a multi-week respiratory muscle training (RMT) program using a handheld breathing device that provides progressive inspiratory and expiratory resistance. Participants also consume a daily standardized dose of beetroot juice concentrate containing dietary nitrate. This combination is expected to enhance breathing muscle strength, vascular function, and exercise tolerance under simulated altitude.
  Interventions: Device: Respiratory Muscle Training (RMT); Dietary Supplement: Dietary Supplement: Beetroot Juice Concentrate
- Respiratory Muscle Training + Placebo (Placebo Comparator): Participants perform the same RMT program as in Arm 1 but consume a placebo beverage that is visually and taste-matched to the nitrate drink but contains no active nitrate. This group allows assessment of the independent effects of respiratory muscle training.
  Interventions: Device: Respiratory Muscle Training (RMT); Dietary Supplement: placebo beverage
- Sham Respiratory Muscle Training + Nitrate Supplementation (Sham Comparator): Participants perform sham RMT with a very low resistance load that does not provide a training stimulus, while consuming the active nitrate beverage daily. This group isolates the independent effect of nitrate supplementation on exercise tolerance under hypoxic conditions.
  Interventions: Device: Sham Respiratory Muscle Training; Dietary Supplement: Dietary Supplement: Beetroot Juice Concentrate
- Sham Respiratory Muscle Training + Placebo (Placebo Comparator): Participants complete sham RMT with minimal breathing resistance and consume a placebo beverage identical in appearance and flavor to the nitrate supplement but containing no active ingredients. This serves as the control condition for comparison with all other intervention groups.
  Interventions: Device: Sham Respiratory Muscle Training; Dietary Supplement: placebo beverage

INTERVENTIONS:
Device: Respiratory Muscle Training (RMT) — Participants perform supervised respiratory muscle training (RMT) using a handheld resistive breathing device designed to strengthen the inspiratory and expiratory muscles. Training sessions are conducted 5 days per week for approximately 4-6 weeks. Each session includes a series of resisted breathing maneuvers with progressively increased load as tolerated. The device is calibrated to maintain a constant pressure threshold to ensure consistent training intensity.
  Other Names: Inspiratory Muscle Training
  Arms: RMT + Nitrate Supplementation; Respiratory Muscle Training + Placebo
Device: Sham Respiratory Muscle Training — Participants use an identical handheld breathing device with minimal resistance, providing no meaningful training stimulus. The training schedule and session duration match those of the active RMT group to maintain participant blinding.
  Arms: Sham Respiratory Muscle Training + Nitrate Supplementation; Sham Respiratory Muscle Training + Placebo
Dietary Supplement: Dietary Supplement: Beetroot Juice Concentrate — Participants consume a standardized dose of concentrated beetroot juice daily for the duration of the training period (approximately 4-6 weeks). The supplement provides a fixed quantity of dietary nitrate known to enhance nitric oxide availability and support vascular and metabolic function during exercise.
  Arms: RMT + Nitrate Supplementation; Sham Respiratory Muscle Training + Nitrate Supplementation
Dietary Supplement: placebo beverage — Participants consume a placebo beverage identical in color, taste, and appearance to the nitrate supplement but containing no active nitrate. The beverage is consumed daily following the same schedule as the active supplement.
  Arms: Respiratory Muscle Training + Placebo; Sham Respiratory Muscle Training + Placebo

SUMMARY:
This study investigates whether respiratory muscle training (RMT) and dietary nitrate supplementation can improve exercise tolerance under simulated moderate altitude conditions. Exposure to reduced oxygen availability at altitude places additional strain on the cardiovascular and respiratory systems, which may limit endurance performance. By combining RMT-designed to strengthen the muscles involved in breathing-with nitrate therapy, which enhances nitric oxide availability and vascular function, this study aims to determine whether these interventions independently or synergistically improve oxygen delivery, reduce physiological strain, and enhance exercise performance. The findings will help identify non-pharmacological strategies to improve physical performance and tolerance to hypoxia in both clinical and operational environments.

DETAILED DESCRIPTION:
This study is designed to test whether two non-drug interventions-respiratory muscle training (RMT) and dietary nitrate supplementation-can improve exercise performance and tolerance when oxygen levels are lower than normal, such as at moderate altitude.

When people exercise in low-oxygen environments, the body must work harder to deliver enough oxygen to the muscles. This can lead to faster fatigue and reduced endurance. Strengthening the breathing muscles and improving blood vessel function may help the body adapt better to these conditions. This study will explore how RMT and nitrate supplementation, either alone or together, affect breathing, blood flow, and exercise capacity.

Why This Study Is Being Done:

Researchers want to find out whether strengthening the breathing muscles through RMT, and increasing nitric oxide in the body through nitrate (found naturally in beetroot juice), can make it easier to exercise when oxygen is limited. Nitric oxide helps widen blood vessels and improve oxygen delivery to muscles. The goal is to learn if these approaches can help healthy adults perform better in low-oxygen conditions and whether combining them produces a greater benefit than using either one alone.

Who Will Participate:

Healthy, recreationally active adults will take part in this study. Participants will not have any known heart, lung, or metabolic disease. They will be randomly assigned to one of four groups:

Breathing training plus nitrate supplement

Breathing training plus placebo

Sham (fake) breathing training plus nitrate supplement

Sham (fake) breathing training plus placebo

What Participants Will Do:

Each participant will complete testing before and after a 4- to 6-week intervention period. During the intervention:

Participants in the RMT group will use a handheld breathing trainer several times per week to strengthen their breathing muscles.

Participants in the nitrate group will drink a small amount of concentrated beetroot juice daily.

Those in the sham groups will use a very low-resistance breathing device or a placebo drink that looks and tastes the same but contains no nitrate.

Before and after training, participants will perform exercise tests on a stationary bicycle both at normal oxygen levels and at simulated altitude inside a controlled environmental chamber. Testing will measure:

How long participants can exercise before becoming fatigued.

Oxygen use (VO₂), heart rate, breathing, and blood pressure during exercise.

Breathing muscle strength and endurance.

Oxygen levels in the blood and muscles.

Study Goals and Measurements:

Researchers will compare how exercise performance and physiological responses change with each treatment. The main goal is to see whether RMT and nitrate supplementation increase exercise tolerance at simulated altitude. Secondary goals include understanding how these interventions affect breathing patterns, oxygen use efficiency, and cardiovascular function during exercise.

Why This Study Matters:

This research will help scientists and health professionals understand how to improve physical performance and resilience when oxygen is limited. The findings could be useful for:

Pilots, military personnel, and athletes who train or work at altitude.

Patients with conditions that make breathing or exercise difficult, such as heart or lung disease.

Future spaceflight or aerospace medicine applications, where oxygen availability can vary.

Safety and Ethics:

All participants will give written informed consent before joining the study. The study has been reviewed and approved by the Institutional Review Board for the Protection of Human Subjects in Research at Embry-Riddle Aeronautical University. All research procedures will follow the ethical principles outlined in the Declaration of Helsinki.

Expected Impact:

The results will show whether combining breathing training with nitrate supplementation can serve as a simple, non-pharmacological strategy to improve tolerance to low-oxygen environments. This could lead to better performance strategies for athletes, aviators, and others who face hypoxic or high-altitude conditions, as well as inform clinical approaches for patients who struggle with exercise intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 40 years old.

Recreationally active (performing ≥3 hours of structured physical activity per week).

Non-smokers for at least the past 6 months.

Free from any known cardiovascular, pulmonary, metabolic, or neuromuscular disease as determined by health screening questionnaire and medical history.

Able to perform cycle ergometer exercise to volitional fatigue.

Willing to abstain from high-nitrate foods and supplements (e.g., beets, spinach, arugula) for 48 hours prior to each testing session.

Able and willing to provide written informed consent and comply with all study procedures.

Exclusion Criteria:

* Diagnosis of or history of heart disease, hypertension, diabetes, or chronic respiratory disorders (e.g., asthma, COPD).

Current use of medications or supplements known to affect cardiovascular, metabolic, or respiratory function (e.g., beta-blockers, nitrates, stimulants).

Smoking, vaping, or tobacco use within the past 6 months.

Known allergy or intolerance to beetroot products or nitrates.

Participation in another interventional research study within the past 30 days.

Pregnant or breastfeeding women.

Any orthopedic or musculoskeletal limitation preventing safe exercise testing.

Failure to meet inclusion criteria or inability to complete familiarization and baseline testing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Tolerance at Simulated Altitude | Baseline to Post-Intervention (approximately 4-6 weeks)
  Exercise tolerance will be measured as the time to exhaustion during a graded cycling exercise test performed under simulated moderate altitude conditions (~2,500-3,000 meters). Tests will be conducted before and after the 4-6 week intervention period. The measure reflects overall improvements in aerobic performance and fatigue resistance following respiratory muscle training, nitrate supplementation, or their combination.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Ferguson, Ph.D., Principal Investigator — Embry-Riddle Aeronautical University
Locations (1):
- Embry-Riddle Aeronautical University, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided